CLINICAL TRIAL: NCT05475483
Title: Phase IIb, Randomized, Double-blind, Placebo-controlled Study in Parallel Groups Assessing the Efficacy and Safety of Two Doses of SOM3355 in Patients Suffering From Huntington's Disease With Choreic Movements
Brief Title: Efficacy and Safety on SOM3355 in Huntington's Disease Chorea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOM Innovation Biotech SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOMCT03; 2021-003453-28 (EudraCT Number)
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Huntington Chorea
Keywords: Huntington; Chorea; SOM3355
MeSH Terms: conditions — Huntington Disease; Chorea | interventions — bevantolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo capsules were administered twice daily (BID) for at least 9 weeks at maintenance dose.
  Interventions: Drug: Placebo capsules
- SOM3355 400 mg/day (Experimental): SOM3355 200 mg capsules were administered twice daily (BID) for at least 9 weeks at maintenance dose.
  Interventions: Drug: SOM3355 200 mg capsules
- SOM3355 600 mg/day (Experimental): SOM3355 300 mg capsules were administered twice daily (BID) for at least 8 weeks at maintenance dose.
  Interventions: Drug: SOM3355 300 mg capsules

INTERVENTIONS:
Drug: Placebo capsules — Treatment was blind for the whole duration of the study.
  Arms: Placebo
Drug: SOM3355 200 mg capsules — Treatment was blind for the whole duration of the study.
  Other Names: Bevantolol hydrochloride
  Arms: SOM3355 400 mg/day
Drug: SOM3355 300 mg capsules — Treatment was blind for the whole duration of the study.
  Other Names: Bevantolol hydrochloride
  Arms: SOM3355 600 mg/day

SUMMARY:
Phase IIb, randomized, double-blind, placebo-controlled study in parallel groups assessing the efficacy and safety of two doses of SOM3355 in patients suffering from Huntington's Disease with choreic movements.

ELIGIBILITY:
Inclusion Criteria: Males or females ≥21 years old, a diagnosis of Huntington's Disease determined by a movement disorders expert and confirmed by a number of HTT gene CAG repeats ≥36, a UHDRS® Total maximal chorea (TMC) score ≥10, and a UHDRS® Total Functional Capacity (TFC) ≥7.

Exclusion Criteria: Onset of HD symptoms prior to age of 21 years (juvenile forms of HD), HD patients presenting rigid akinesia, and use of other VMAT2 inhibitors such as tetrabenazine, deutetrabenazine, or valbenazine, or other antichoreic treatment such as any neuroleptic, or amantadine, memantine, riluzole.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- France (5):
  - Centre Hospitalier Universitaire Angers, Angers
  - CHU Hôpital Henri Mondor (APHP), Créteil
  - Hôpital Roger Salengro - CHU Lille, Lille
  - Hopital de Hautepierre, Strasbourg
  - Hôpital Purpan - CHU Toulouse, Toulouse
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - George Huntington Institut, Münster
  - Kbo-Isar-Amper-Klinikum Taufkirchen, Taufkirchen
  - Hospital of University of Ulm, Ulm
- Italy (4):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - IRCCS Casa Sollievo della Sofferenza, Roma
  - Sant'Andrea University Hospital, Roma
- Poland (2):
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - Indywidualna Praktyka Lekarska Daniel Zielonka, Poznan
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Ramón y Cajal, Madrid
- Universitaetsspital Bern - Inselspital, Bern, Switzerland
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust Addenbrooke's Hospital, Cambridge
  - NIHR Wellcome Trust Manchester Clinical Research Facility, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: SOM Biotech website — http://www.sombiotech.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 139 patients with Huntington's disease were randomized and treated between August 2022 and April 2024 at 23 sites in 7 European countries.
Period: Overall Study
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day
Started | 48 | 41 | 50
Completed | 41 | 36 | 41
Not Completed | 7 | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day | Total
Number analyzed (Participants) | 48 | 41 | 50 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 32 | 45 | 120
  >=65 years | 5 | 9 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.65 (10.46) | 52.51 (12.39) | 51.34 (12.12) | 51.79 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 17 | 21 | 66
  Male | 20 | 24 | 29 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: White | 48 | 39 | 48 | 135
  Ethnic Origin: African (North) | 0 | 1 | 1 | 2
  Ethnic Origin: Latino | 0 | 1 | 0 | 1
  Ethnic Origin: Other (in France) | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Poland | 8 | 9 | 9 | 26
  Italy | 5 | 6 | 8 | 19
  United Kingdom | 7 | 4 | 7 | 18
  France | 7 | 2 | 6 | 15
  Switzerland | 2 | 1 | 2 | 5
  Germany | 7 | 7 | 7 | 21
  Spain | 12 | 12 | 11 | 35
Use of Neuroleptics [Count of Participants; unit: Participants] — Antipsychotic drugs (excluding haloperidol, pimozide, and tiapride) prescribed to treat behaviour disorders at a stable dose for at least 3 months before entering the study.
  Participants
    Yes | 6 | 5 | 6 | 17
    No | 42 | 36 | 44 | 122
Total Maximal Chorea (TMC) score [Mean (Standard Deviation); unit: units on a scale] — The TMC is part of the motor assessment of the Unified Huntington's Disease Rating Scale (UHDRS) and measures chorea in 7 different body parts, including the face, oral-buccal-lingual region, trunk, and each limb independently. The TMC score is the sum of the individual scores, ranging from 0 to 28. Lower values in the TMC score represent less chorea symptoms and a better outcome.
  units on a scale | 12.80 (2.58) | 12.74 (2.93) | 13.23 (2.84) | 12.94 (2.77)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Maximal Chorea (TMC) Score of the UHDRS® for Subjects Not Taking Neuroleptics During the Trial (mITT - N=122)
Description: Pre-defined analysis of the primary efficacy endpoint (change in TMC score from baseline to the end of maintenance dose) performed with the 122 subjects of the mITT not taking neuroleptics during the trial.
  The TMC is part of the motor assessment of the Unified Huntington's Disease Rating Scale (UHDRS) and measures chorea in 7 different body parts, including the face, oral-buccal-lingual region, trunk, and each limb independently. The TMC score is the sum of the individual scores, ranging from 0 to 28. A decrease in TMC scores indicates improvement in chorea symptoms.
Time Frame: From baseline to end of maintenance dose (10 weeks of treatment).
Population: 122 subjects of the mITT not taking neuroleptics during the trial. The modified Intention-to-Treat (mITT) population comprises all patients randomized to a treatment arm who received at least one dose of study drug and had at least one post-baseline assessment of the TMC score (N=139).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day
Number analyzed (Participants) | 42 | 36 | 44
units on a scale | -2.19 [-3.07 to -1.32] | -2.42 [-3.32 to -1.51] | -3.46 [-4.35 to -2.58]
Statistical Analysis 1: Comparison: Placebo vs SOM3355 600 mg/Day; Test type: Other; p = 0.045, Mixed Models Analysis; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-2.51 to -0.03]

2. Secondary Outcome: Change in the Clinical Global Impression (CGI) (mITT - N=139)
Description: The key secondary endpoint was the Clinical Global Impression of Change (CGI-C) at Visit 5 (week 10). The key secondary efficacy analysis was conducted on the mITT Population, including 139 subjects. Subjects with a score of 1 (Very much improved), 2 (Much improved), or 3 (Minimally improved) were defined as "Improved", and patients with a score of 4 (No change), 5 (Worse), 6 (Much worse), and 7 (Very much worse) were defined as "Not Improved".
Time Frame: From baseline to end of maintenance dose (10 weeks of treatment).
Population: Modified Intention-to-Treat (mITT) population included all patients randomized to a treatment arm, who received at least one dose of study drug and had at least one post-baseline assessment of the TMC score.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day
Number analyzed (Participants) | 41 | 37 | 41
Participants
  Improved | 15 | 26 | 23
  Not Improved | 26 | 11 | 18
Statistical Analysis 1: Comparison: Placebo vs SOM3355 600 mg/Day; Test type: Other; p = 0.078, Regression, Logistic; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.91 to 5.37]

3. Secondary Outcome: Change in the Patient Global Impression (PGI) (mITT - N=139)
Description: Another relevant secondary endpoint was the Patient Global Impression of Change (PGI-C) at Visit 5 (week 10). The efficacy analysis was conducted on the mITT Population, including 139 subjects. Subjects with a score of 1 (Very much improved), 2 (Much improved), or 3 (Minimally improved) were defined as "Improved", and patients with a score of 4 (No change), 5 (Worse), 6 (Much worse), and 7 (Very much worse) were defined as "Not Improved".
Time Frame: From baseline to end of maintenance dose (10 weeks of treatment).
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day
Number analyzed (Participants) | 41 | 37 | 40
Participants
  Improved | 20 | 25 | 26
  Not Improved | 21 | 12 | 14
Statistical Analysis 1: Comparison: Placebo vs SOM3355 600 mg/Day; Test type: Other; p = 0.143, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.80 to 4.76]

4. Post Hoc Outcome: Change in Total Maximal Chorea (TMC) Score for Subjects Not Taking Neuroleptics and With Mean Baseline TMC Score >12 (mITT - N=57)
Description: Post-hoc analysis of the primary efficacy endpoint (change in TMC score from baseline to the end of maintenance dose) was performed in 57 subjects of the mITT not taking neuroleptics during the trial and with a mean baseline TMC score >12. The TMC is part of the motor assessment of the Unified Huntington's Disease Rating Scale (UHDRS) and measures chorea in 7 different body parts, including the face, oral-buccal-lingual region, trunk, and each limb independently. The TMC score is the sum of the individual scores, ranging from 0 to 28. A decrease in TMC scores indicates improvement in chorea symptoms.
Time Frame: From baseline to end of maintenance dose (10 weeks of treatment).
Population: 57 subjects of the mITT not taking neuroleptics during the trial and with a mean baseline TMC score >12.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day
Number analyzed (Participants) | 21 | 14 | 22
units on a scale | -2.43 [-3.57 to -1.28] | -2.76 [-4.20 to -1.32] | -4.21 [-5.36 to -3.06]
Statistical Analysis 1: Comparison: Placebo vs SOM3355 600 mg/Day; Test type: Other; p = 0.032, Mixed Models Analysis; Mean Difference (Final Values) = -1.78, 95% CI 2-sided [-3.40 to -0.16]

ADVERSE EVENTS:
Time Frame: From Baseline (visit 1) until End of Study visit (up to 13 weeks of treatment).
Arm/Group | Placebo | SOM3355 400 mg/Day | SOM3355 600 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/41 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/48 | 1/41 | 1/50
Other Adverse Events (participants affected / at risk) | 10/48 | 15/41 | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=48) | SOM3355 400 mg/Day (N=41) | SOM3355 600 mg/Day (N=50)
Syncope (overdose) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=48) | SOM3355 400 mg/Day (N=41) | SOM3355 600 mg/Day (N=50)
Fall (Injury, poisoning and procedural complications) | 2 (5) | 3 (6) | 4 (7)
Bradycardia (Vascular disorders) | 0 (0) | 2 (2) | 6 (7)
Somnolence (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (6) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05475483/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT05475483/SAP_001.pdf